CLINICAL TRIAL: NCT02656407
Title: Doppler Ultrasonore Ultrasensible Peropératoire du Cerveau - Vers Une Aide Temps Reel à la Cartographie Corticale Fonctionnelle
Brief Title: Intraoperative Functional Ultrasound
Acronym: FUSIMAGINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: C14-66; 2015-A00661-48 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2015-12-17; First posted 2016-01-15 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2021-08

CONDITIONS: Brain Tumor; Brain Lesion
Keywords: Functional Ultrasound; Intraoperative; Brain; Doppler; Ultrasound
MeSH Terms: conditions — Brain Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasensitive Doppler (Experimental): Intraoperative ultrasensitive Doppler acquisitions by using an ultrasound device for functional area detection
  Interventions: Device: Ultrasound device

INTERVENTIONS:
Device: Ultrasound device — Ultrasensitive Doppler acquisition obtained with the Aixplorer ultrasound device

SUMMARY:
A wide spectrum of methods is used to image brain activation in vivo. It can be directly detected by neurons electrical activity imaging (cortical simulation mapping, calcium imaging, voltage sensitive dyes) or indirectly by imaging hemodynamic changes induced by the neurovascular coupling in the vessels surrounding the activated neurons (intrinsic optical imaging, photoacoustic imaging, positron emission tomography (PET), functional magnetic resonance imaging (fMRI)).

Ultrasound as the potential to complement these functional imaging techniques at low cost. Ultrasound imaging can do real-time in-depth imaging of brain. However, its use to imaging of major vessels has been limited until now due to its poor sensitivity. To overcome this limitation functional ultrasound (fUS) was developed in Institut Langevin since 2011. This technique enables high spatio-temporal resolution imaging of whole-brain microvasculature dynamics in response to brain activation without the need of contrast agent.

This fUS method relies on a new power Doppler imaging sequence sensitive enough to detect blood flow in most of cerebral vessels (arterioles, big venules and larger vessels). Repeating the acquisition of such ultrasensitive Doppler images over time enables to follow flow dynamics in such vessels modulated by local neuronal activity.

Applied to the rat brain, fUS was proved able to map brain activation at high spatiotemporal resolution and high signal to noise ratio. The aim of this study is now to apply fUS on human brain in intraoperative condition.

The main objective of this study is to find activation maps through intraoperative ultrasensitive Doppler compared to gold standard cortical simulation mapping and functional MRI.

Secondly the investigators want to test sensitivity of this new Doppler mode. fUS method will be used for different types of stimuli and intensity and the investigators will do some control acquisitions. Blood vessel density observed with a conventional Doppler will be compared to the one measured with the ultrasensitive Doppler to prove that this new Doppler mode enhance micro vessel visualization.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, adults ( > 18 years old)
* Participants who have to undergo brain surgery, awake or under general anesthesia, for tumor or lesion resection (all types of tumors and lesions, cortical or subcortical), with programmed intraoperative ultrasound and cortical simulation mapping.
* Consent form signed by the patient after being informed (written and oral) of the research protocol.
* Patient affiliate to the social welfare system

Exclusion Criteria:

* Minors ( < 18 years old)
* Pregnant, parturient or breastfeeding women
* Protected persons, under guardianship, or under any administrative or legal right and liberty revocation procedure
* Patient without affiliation to the social welfare system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Activation maps through intraoperative ultrasensitive Doppler compared to gold standards cortical simulation mapping and functional MRI | During the surgery

SECONDARY OUTCOMES:
Sensitivity test of the new Doppler mode | During surgery
  fUS method will be tested for different types of stimuli and intensity and the investigators will do some control acquisitions.
In depth micro vessel localization | During surgery
  Blood vessel density observed with a conventional Doppler will be compared to the one measured with the ultrasensitive Doppler.

CONTACTS AND LOCATIONS:
Overall Officials: Dorian Chauvet, MD, Principal Investigator — Neurosurgery department
Locations (1):
- Pitié Salpetriere Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Imbault M, Chauvet D, Gennisson JL, Capelle L, Tanter M. Intraoperative Functional Ultrasound Imaging of Human Brain Activity. Sci Rep. 2017 Aug 4;7(1):7304. doi: 10.1038/s41598-017-06474-8. PMID 28779069
- [Background] Demene C, Deffieux T, Pernot M, Osmanski BF, Biran V, Gennisson JL, Sieu LA, Bergel A, Franqui S, Correas JM, Cohen I, Baud O, Tanter M. Spatiotemporal Clutter Filtering of Ultrafast Ultrasound Data Highly Increases Doppler and fUltrasound Sensitivity. IEEE Trans Med Imaging. 2015 Nov;34(11):2271-85. doi: 10.1109/TMI.2015.2428634. Epub 2015 Apr 30. PMID 25955583